CLINICAL TRIAL: NCT02924168
Title: Effect of Radial Shock Waves for the Treatment of Upper Limb Functional Disability in Stroke Sequelae
Brief Title: Radial Shock Waves for Functional Disability in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Imamura (Other)
Responsible Party: Sponsor-Investigator, Marta Imamura, MD PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19109813.1.0000.0068
Record Dates: First submitted 2016-09-29; First posted 2016-10-05 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Radial Shockwave (Experimental): Every patient will receive 5,000 continuous pulses per treatment session, at 3.5 to 4 bar air pressure (resulting in an energy flux density [EFD] of approximately 0.07 mJ/mm2) and at 15Hz frequency. A total of 4 sessions will be performed.
  Interventions: Device: Active Radial Shockwave
- Sham Radial Shockwave (Sham Comparator): Every patient will receive 5,000 continuous pulses per treatment session, without air pressure (resulting in no EFD) and at 15Hz frequency. A total of 4 sessions will be performed.
  Interventions: Device: Sham Radial Shockwave

INTERVENTIONS:
Device: Active Radial Shockwave — Four weekly sessions of active radial shockwave treatment.
  Arms: Active Radial Shockwave
Device: Sham Radial Shockwave — Four weekly sessions of sham radial shockwave treatment.
  Arms: Sham Radial Shockwave

SUMMARY:
This is a double blind randomized clinical trial to evaluate the effect of radial shock waves on functional recovery of the upper limb of patients with sequelae of ischemic strokes in the territory of the middle cerebral artery. A total of 20 patients will be enrolled and will undergo motor, functional and cortical excitability evaluations before and after four weekly sessions of radial shockwaves. 5,000 pulses with a frequency of 15 Hz and 3.5 to 4 bar of air pressure will be applied to the active group, resulting in an energy flux density (EFD) of approximately 0.07 mJ/mm2. The sham group will receive identical treatment, except for the fact that no energy flux will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis: Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) scan indicating Stroke in the territory of the middle cerebral artery;
* 6 to 24 months after stroke date;
* Stability observed in clinical medical evaluation
* Granting of written informed consent to participate in the study

Exclusion Criteria:

* Individuals with a score lower than 24 on the Mini-mental test;
* Previously documented strokes
* Pregnancy
* Patients treated with botulinum toxin, phenol, alcohol or previous surgeries six months before entering the study
* Bone diseases, pre-existing joint damage, and deformities affecting the patient in a way to interfere with implementation of the proposed therapy
* Psycho-affective disorder that prevents adherence
* Joint pain that occurs within the movement range of therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Change from baseline to 8 weeks
  Mean change in Fugl Meyer Assessment score after four sessions of Radial Shockwave Therapy (RSWT) as compared to baseline.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline, one and two months
  Multiple changes in VAS
Esthesiometry - Von Frey Scale | Baseline, one and two months
  Multiple changes in Von Frey Scale
Upper Limb Modified Ashworth Scale (MAS) | Baseline, one week, two weeks, three weeks, four weeks and two months
  Multiple changes in MAS
Fugl-Meyer Assessment | Baseline and two months
  Changes in Fugl-Meyer Assessment compared to baseline
Medical Research Council scale (MRC) | Baseline, one and two months
  Multiple changes in MRC scale
Hand grip | Baseline, one and two months
  Multiple changes in Hand grip
Change in fine motor function measured with Finger Tapping (FT) | Baseline, one and two months
  Multiple changes in FT
Jebsen-Taylor Hand Function Test (JTHFT) | Baseline, one and two months
  Multiple changes in JTHFT
Purdue Pegboard Test (PPBT) | Baseline, one and two months
  Multiple changes in PPBT
Robotic kinematic evaluation (RKE) | Baseline, one and two months
  Multiple changes in RKE
Corticospinal excitability measures with transcranial magnetic stimulation (TMS) | Baseline, one and two months
  Multiple changes in Corticospinal excitability
Pinch strength testing | Baseline, one and two months
  Pinch strength testing

OTHER OUTCOMES:
Adverse Events (AE) | Weekly for two months
  Accountability of occurences of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD, Principal Investigator — Instituto de Medicina Física e Reabilitação HCFMUSP
Locations (1):
- Instituto de Medicina Fisica e Reabilitacao HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No